CLINICAL TRIAL: NCT06808438
Title: Research on Precision Individualized Mechanical Ventilation Strategies for ARDS Guided by Electrical Impedance Tomography Monitoring and Evaluation of the Differences in Ventilation and Perfusion Distribution
Brief Title: Incremental and Decremental PEEP Titration by Diverse Strategies in Subjects with ARDS: a Prospective Physiological Study
Acronym: ARDS，PEEP
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhou Yongfang, Chief respiratory therapist, Sichuan University
Other Study IDs: PEEP Titration; 2022YFC2504403 (Other Grant/Funding Number: National Key R＆D Program of China)
Record Dates: First submitted 2024-12-05; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-12

CONDITIONS: ARDS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Esophageal pressure catheter — Esophageal pressure was monitored with an esophageal pressure catheter

SUMMARY:
The investigators conducted a prospective physiological observation study on ARDS population, described their physiological and EIT indexes with various PEEP titration methods, and also compared and analyzed those indexes to determine whether there were differences among various PEEP titration methods.The objective of this study was to explore and uncover the physiological differences in response to optimal PEEP in different ways，and analyzed the correlation of the optimal PEEP in these different ways.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanical ventilated patients in ICU within 48 hours
* Be over 18 years old
* With moderate-severe ARDS (PaO2 /FIO2 ,200 mm Hg)

Exclusion Criteria:

* Severe chronic obstructive pulmonary diseases
* Pulmonary bulla(>1CM) or pneumothorax or pneumomediastinum or subcutaneous emphysema
* Pregnancy
* BMI≥35kg/m2
* Suspected pulmonary vascular hemorrhage
* Disturbance of consciousness or intracranial hypertension
* Severe cardiac dysfunction (New York Heart Association Class III or IV, acute -Coronary syndrome or persistent ventricular tachyarrhythmia), cardiogenic shock or after major cardiac surgery
* Hemodynamic instability (i.e., mean arterial pressure [MAP]<60 mm Hg despite vasopressor use
* The medical team considering short periods of high pressure to be unsafe
* Contraindications for placement of esophageal pressure catheters (e.g., esophageal varix or fracture of skull base)
* Contraindications for EIT monitoring (including pacemaker, or cutaneous diseases which limiting electrode placement)
* Agonal stage or end-stages of diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ntubated and mechanical ventilated patients over 18 years with moderate-severe ARDS (PaO2 /FIO2 ,200 mm Hg) admitted to the ICU within 48 hours were enrolled from October 2022 to July 2024.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
the value of set PEEP | through study completion, an average of 1 year
  Select the optimal PEEP value according to different ways

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No